CLINICAL TRIAL: NCT04973202
Title: Portrayal of Hospital Alcohol Detoxifications and Factors Associated With Longer or Ulterior Hospitalizations in France From 2011 to 2020
Brief Title: Portrayal of Hospital Alcohol Detoxification in France
Acronym: Alcostop
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0456
Record Dates: First submitted 2021-07-06; First posted 2021-07-22 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Alcohol Use Disorder; Addiction; Alcohol Withdrawal Syndrome
Keywords: National portrayal of hospital alcohol detoxification in France; Rehabilitation in France; Alcohol in French hospitals and clinics; Alcohol detoxification
MeSH Terms: conditions — Alcoholism; Behavior, Addictive | interventions — Ethanol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Inpatients for alcohol detoxifications: French patients who were hospitalized for alcohol detoxification from 2011 to 2020
  Interventions: Other: Stay for alcohol detoxification

INTERVENTIONS:
Other: Stay for alcohol detoxification — Stay for alcohol detoxification : routine care.

SUMMARY:
Even if hospital alcohol detoxifications are frequent in France, their caracteristicscharacteristics remain unknown. The investigators aim to describe the clinical and paraclinical caracteristicscharacteristics of their patients, their length and geographical repartition, etc… The investigators also aim to evaluate factors associated with longer stays or ulterior re-hospitalization for the same reason. Finally, The investigators aim to compare the stays by facility type.

DETAILED DESCRIPTION:
Context:

In France, the consequences of excessive alcohol use are one of the primary reasons for hospitalization. When stopping the substance, patients with an alcohol use disorder can suffer from a potentially fatal alcohol withdrawal syndrome. To mitigate these risks, a withdrawal under medical supervision is possible, either in an outpatient setting or in hospital, where the detoxification can be programmed or imposed. In the course of an alcohol dependent patient's life, re-drinking is not exceptional and the patient may undergo several withdrawals during his or her life.

Psychiatric pathologies, especially anxiety and depression, are more frequent in these patients than in the rest of the population, just as can be somatic pathologies.e. Withdrawal accidents, represented by comital seizures and delirium tremens, can be critical.

In hospital detoxifications, studies do not show any benefit in continuing the stay beyond 10 days, except in the case of somatic or psychiatric complication. However, little information is available on the average length of stay for hospital alcohol detoxification.

Although alcohol dependence issues are very frequent and the resulting withdrawals are relatively common and associated with numerous comorbidities, little data exists at a national level in France.

The aim of this study is to describe these hospital detoxifications: course, duration, frequency and clinical and paraclinical characteristics of the patients. We also wish to analyze which characteristics are associated with longer stays or re-hospitalization and to compare the care according to the facility type.

Objectives:

Main:

- To describe the clinical, paraclinical, and stay characteristics of hospital alcohol detoxification in France

Secondary:

* To describe the regional distribution of hospital alcohol detoxification
* To evaluate whether certain clinical characteristics are associated with a longer hospital stays
* To evaluate whether certain clinical characteristics are associated with subsequent re-hospitalization for the same reason
* To compare the characteristics of patient stays by type of facility

Methods:

In this descriptive observational study using pre-existing data accessed via the PMSI (Programme de Médicalisation des Systèmes d'Information), we will use all hospital stays from 2011 to 2020 for alcohol detoxification in France, both in public and private settings.

For each hospital stay will be collected the length, the antecedents of hospital alcohol detoxification, clinical and psychiatric comorbidities, withdrawals complication, alcohol use complication, further examinations.

We will describe the stays using median and quartiles for continuous variables and number and percentage for dichotomous variables. For secondary objectives, we will use a multivariate linear regression model if the length of stay is normal, an ordinal regression model otherwise. The characteristics of the stays will be compared regarding the type of facility using univariate comparative tests: Chi² or Fisher for dichotomous variables and Student or Mann-Whitney for continuous variables.

ELIGIBILITY:
Inclusion criteria:

Inclusion criteria:

* French patients of at least 18 years old
* Inpatients of a public or private care facility for alcohol detoxification
* From 01/01/2011 to 12/31/2020
* In a medical or psychiatric hospital

Exclusion criteria:

- age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: French patients hospitalized for alcohol detoxification from 2011 to 2020
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
description of age | day 1 (At hospital inclusion)
  Age at admission (in years), calculated by the difference of the year of admission and the year of birth through the PMSI.
description of sex | day 1 (At hospital inclusion)
  Sex collected through the PMSI.

SECONDARY OUTCOMES:
description of geographic code | day 1 (At hospital inclusion)
  Sex collected through the PMSI.
description of CMU-C | day 1 (At hospital inclusion)
  CMU-C (universal complementary health insurance, collected through the PMSI.
Length of stay | During the stay (day 1 - day 15)
  Length of stay (in days), calculated by the difference between the discharge date and the entry date, collected through the PMSI.
Care establishment | During the stay (day 1 - day 15)
  Name and type of the care establishment, collected through the PMSI.
Number of previous hospital detoxification stays in the studied period | During the stay (day 1 - day 15)
  Number of previous hospital detoxification stays in the studied period, collected through the PMSI.
Psychiatric comorbidities | During the stay (day 1 - day 15)
  Psychiatric comorbidities (Major depression episode, anxiety, psychotic trouble, personality diseases), collected through the PMSI.
Withdrawal complication | During the stay (day 1 - day 15)
  Withdrawal complications (delirium tremens, comitial seizures), collected through the PMSI.
Further examination | During the stay (day 1 - day 15)
  Further examination (biology, imagery, etc…), collected through the PMSI.
Re-hospitalization for same reason | day 1
  For each patient, and each stay, we will evaluate if the patient had an ulterior re-hospitalization for alcohol withdrawal. Collected through the PMSI.

CONTACTS AND LOCATIONS:
Overall Officials: Lionel MOULIS, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC